CLINICAL TRIAL: NCT01544972
Title: Serum Level Measurement of Oral Paracetamol and Oral Ibuprofen
Brief Title: Serum Level Measurement of Oral Paracetamol and Oral Ibuprofen for Patent Ductus Arteriosus Treatment in Preterm Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Sadik Yurttutan, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZTB170212
Record Dates: First submitted 2012-02-22; First posted 2012-03-06 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent Ductus Arteriosus; Paracetamol; Ibuprofen; Serum levels; Preterm infant
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral paracetamol (Active Comparator): Patients will receive oral paracetamol 15 mg/kg per dose every 6 hours for 3 days
  Interventions: Drug: Oral paracetamol
- Oral ibuprofen (Active Comparator): Patients will receive oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h.
  Interventions: Drug: Oral ibuprofen

INTERVENTIONS:
Drug: Oral paracetamol — Patients will receive oral paracetamol 15 mg/kg per dose every 6 hours.
  Other Names: Calpol
  Arms: Oral paracetamol
Drug: Oral ibuprofen — Patients will receive oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h.
  Other Names: Pedifen
  Arms: Oral ibuprofen

SUMMARY:
The purpose of this study is to determine oral paracetamol and ibuprofen efficacy and safety in relation to serum levels in closure of patent ductus arteriosus in preterm infants.

DETAILED DESCRIPTION:
To determine oral paracetamol and ibuprofen efficacy and safety in relation to serum levels in closure of patent ductus arteriosus in preterm infants.

Eighty preterm infants with patent ductus arteriosus will be enrolled in this prospective-randomized study. Patients will receive oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h or oral paracetamol 15 mg/kg per dose every 6 hours for 3 days.

One of the following echocardiographic criteria of a duct size > 1.5 mm, a left atrium-to-aorta ratio > 1.5, left-to-right shunting of blood, end diastolic reversal of blood flow in the aorta, or poor cardiac function in addition signs of patent ductus arteriosis determined the need of treatment.

Three consecutive blood sample from infants for 3 days before dose application of drugs(ibuprofen and paracetamol will be obtained.

The relation of pharmacokinetics of drugs to drug response will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Birth weight below 1250 gram
* Diagnosed patent ductus arteriosus by Echocardiographic examination

Exclusion Criteria:

* Accompanied other congenital cardiac anomalies
* Severe thrombocytopenia < 60.000
* Severe intracranial bleeding (Grade III - IV)
* Intestinal abnormality and necrotising enterocolitis

Ages: 2 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To detection of safe and effective serum levels of paracetamol and ibuprofen in preterm infants treated for PDA | up to 6 months
  The measurement of Serum levels of Paracetamol and Ibuprofen in preterm infants treated with Oral Paracetamol and Oral Ibuprofen.
  To determine of effective serum levels of paracetamol and ibuprofen for treatment of patent ductus arteriosus in preterm infants.
  In normally, effective and safely dose of NSAIDs for treatment of PDA are exactly unknown. Therefore we will detected cut-off serum levels for effective, safely and hazardous.

CONTACTS AND LOCATIONS:
Overall Officials: Sadık Yurttutan, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Division of Neonatology, Ankara, Turkey (Türkiye)